CLINICAL TRIAL: NCT04566497
Title: Assessment in a Randomized Controlled Trial of Adverse Outcome in Asymptomatic Patients With Prior Coronary Revascularization Who Have a Systematic Stress Testing Strategy Or a Non-testing Strategy During Long-term Follow-up.
Brief Title: Assessment of Adverse Outcome in Asymptomatic Patients With Prior Coronary Revascularization Who Have a Systematic Stress Testing Strategy Or a Non-testing Strategy During Long-term Follow-up.
Acronym: ARCACHON
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P170908J
Record Dates: First submitted 2020-08-31; First posted 2020-09-28 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention; Coronary Artery Bypass Grafting
Keywords: Stress testing; Myocardial ischemia; Coronary artery disease; coronary revascularization
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia | interventions — 26S proteasome non-ATPase regulatory subunit 13; Exercise Test; DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): no systematic stress testing during follow-up
  Interventions: Other: No stress testing
- Active Comparator (Active Comparator): systematic annual stress testing during follow-up
  Interventions: Procedure: stress testing

INTERVENTIONS:
Other: No stress testing — No stress testing during the patient follow up (up to 48 months) if the patient remains asymptomatic
  Other Names: Arm1
  Arms: Experimental
Procedure: stress testing — Systematic annual stress testing during the patient follow up (up to 48 months)
  Other Names: Arm 2
  Arms: Active Comparator

SUMMARY:
Due to the lack of randomized controlled trials, the best follow-up strategy of asymptomatic patients after coronary artery revascularization is controversial. A systematic screening of silent myocardial ischemia may help prevent a major acute cardiac event. However, systematic screening strategy is costly and there is currently no evidence that repeated revascularization improve survival. Moreover, stress testing per se or additional procedures which can be performed with regard of stress testing results can cause unexpected complications.

ARCACHON is a national, multicenter, randomized, open label trial, that will evaluate the non-inferiority of a clinical follow-up as compared to a systematic stress testing strategy after coronary revascularization.

DETAILED DESCRIPTION:
Coronary artery revascularization is commonly used for the management strategy of patients with coronary artery disease (CAD).

In the following years after revascularization, the current guidelines recommend evaluation with stress tests when patients are symptomatic. Due to the lack of randomized trials, the evaluation of asymptomatic patients is controversial and accordingly there is a wide variation in routine follow-up strategies in these patients. A systematic screening of silent myocardial ischemia may help prevent a major acute cardiac event. However, systematic screening strategy is costly and there is currently no evidence that repeated revascularization improve survival We hypothesized that clinical follow-up alone would be non-inferior to systematic stress testing screening strategy during follow-up of asymptomatic CAD patients with prior coronary revascularization.

The primary objective of ARCACHON trial is to demonstrate the non-inferiority of a strategy of clinical follow-up (without non-invasive stress testing) in asymptomatic patients with a history of coronary revascularization compared to a strategy of systematic screening for myocardial ischemia using non-invasive stress testing by the primary endpoint as the composite of: all-cause death, myocardial infarction, stroke or any cardiovascular event leading to unplanned hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Prior coronary revascularization (PCI or CABG) at any time before randomization.
2. Asymptomatic at the time of randomization (defined as a Canadian Cardiovascular Society score ≤ 1, stable on the current medical treatment).
3. Patient affiliated to Social Security
4. Informed, written consent from the patient

Exclusion Criteria:

1. Age < 18years
2. Any acute coronary syndrome in the previous 3 months
3. Symptoms suggestive of angina pectoris at the time of randomization:

   * Angina is characterized by ischemic chest pain occurring on exertion or stress relieved by rest and/or nitroglycerine.
   * Angina equivalents are defined as dyspnea, fatigue, or diaphoresis on exertion evaluated by the principal investigator as abnormal and attributable to myocardial ischemia.
4. Any severe valvular disease
5. Prior heart transplantation
6. Class III or IV symptomatic heart failure (NYHA classification).
7. Persons whose occupations impact on public safety (e.g. airline pilots, lorry or bus drivers) in whom systematic stress testing could be required for medico-legal reasons
8. Malignancies and other comorbid conditions with a life expectancy < 2 years
9. Pregnancy or nursing women
10. Women of childbearing age without effective birth control or intention to become pregnant during the course of the trial
11. Simultaneous enrollment in an interventional clinical trial and interventional research with minimal risks and burden
12. Inability to sign an informed consent. Patient under legal protection (guardianship, curatorship) or mental condition (psychiatric or organ cerebral disease) rendering the subject unable to understand the nature, scope, and possible consequences of the trial or mental retardation or language barrier such that the patient is unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2664 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
demonstrate the non-inferiority of a strategy of clinical follow-up | minimum 24 months to 48 months
  The primary outcomes measured at longest follow-up (minimum 24 months) the number of All-cause death in each arm
demonstrate the non-inferiority of a strategy of clinical follow-up | minimum 24 months to 48 months
  The primary outcomes measured at longest follow-up (minimum 24 months) is the number of Myocardial infarction in each arm
demonstrate the non-inferiority of a strategy of clinical follow-up | minimum 24 months to 48 months
  The primary outcomes measured at longest follow-up (minimum 24 months) is the number of Stroke in each arm
  hospitalization.
demonstrate the non-inferiority of a strategy of clinical follow-up | minimum 24 months to 48 months
  The primary outcomes measured at longest follow-up (minimum 24 months) is the number of any cardiovascular event leading to unplanned hospitalization in each arm

SECONDARY OUTCOMES:
compare the clinical follow-up strategy to a systematic screening of myocardial ischemia | minimum 24 months to 48 months
  Hierarchical assessment of the following criteria at longest follow-up (minimum 24 months) All-cause death, myocardial infarction
compare the clinical follow-up strategy to a systematic screening of myocardial ischemia | minimum 24 months to 48 months
  Hierarchical assessment of the following criteria at longest follow-up (minimum 24 months): Angina control per Seattle Angina Questionnaire
compare the clinical follow-up strategy to a systematic screening of myocardial ischemia | minimum 24 months to 48 months
  Hierarchical assessment of the following criteria at longest follow-up (minimum 24 months): Quality of life in each arm
compare the clinical follow-up strategy to a systematic screening of myocardial ischemia | minimum 24 months to 48 months
  Hierarchical assessment of the following criteria at longest follow-up (minimum 24 months): Urgent or unscheduled revascularizations in each arm
compare the clinical follow-up strategy to a systematic screening of myocardial ischemia | minimum 24 months to 48 months
  Hierarchical assessment of the following criteria at longest follow-up (minimum 24 months): Any cardiovascular event leading to unplanned hospitalization in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Nadjib Hammoudi, MD PHD, Principal Investigator — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS
Locations (1):
- Pitie salpetriere, Paris, France

IPD SHARING:
Plan to Share IPD: No